CLINICAL TRIAL: NCT00914316
Title: Supervised Treadmill Exercise and Ranolazine for Intermittent Claudication of Lower Extremities. THE STERILE TRIAL.
Brief Title: Supervised Treadmill Exercise and Ranolazine for Intermittent Claudication of Lower Extremities
Acronym: STERILE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Corewell Health East (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2009-051
Record Dates: First submitted 2009-06-02; First posted 2009-06-04 (Estimated); Results first posted 2017-08-09 (Actual); Last update posted 2017-08-09 (Actual); Status verified 2017-06

CONDITIONS: Peripheral Arterial Disease
Keywords: Lower leg claudication; Poor circulation of the leg muscles; Cramping or discomfort in the lower legs; Lower leg pain; PAD (Peripheral arterial disease)
MeSH Terms: conditions — Peripheral Arterial Disease; Spasm | interventions — Ranolazine; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Phase 1-Ranolazine, Phase 2-Ranolazine (Active Comparator): This group will participate in the Phase 1 -12 week supervised exercise program and will additionally receive ranolazine 1000 mg orally, twice daily, by mouth. In Phase 2, the group will exercise independently and also receive ranolazine 1000 mg orally twice daily by mouth.
  Interventions: Drug: Ranolazine
- Phase 1 -Ranolazine, Phase 2 -Placebo (Active Comparator): This group will participate in the Phase 1 -12 week supervised exercise program and will additionally receive ranolazine 1000 mg orally, twice daily, by mouth. In Phase 2, the group will exercise independently and will receive a sugar pill in place of the study drug.
  Interventions: Drug: Ranolazine; Drug: Placebo
- Phase 1 -Placebo, Phase 2 -Ranolazine (Active Comparator): This group will participate in the Phase 1 -12 week supervised exercise regimen and will receive a sugar pill in place of the study drug. In Phase 2, the group will exercise independently and also receive ranolazine 1000 mg orally twice daily by mouth.
  Interventions: Drug: Ranolazine; Drug: Placebo
- Phase 1 -Placebo, Phase 2 -Placebo (Placebo Comparator): This group will participate in the Phase 1 -12 week supervised exercise regimen and will receive a sugar pill in place of the study drug. In Phase 2, the group will exercise independently and will receive a sugar pill in place of the study drug.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ranolazine — Ranolazine, 1000 mg, capsule, twice daily, by mouth.
  Other Names: Ranexa
  Arms: Phase 1 -Placebo, Phase 2 -Ranolazine; Phase 1 -Ranolazine, Phase 2 -Placebo; Phase 1-Ranolazine, Phase 2-Ranolazine
Drug: Placebo — twice daily
  Other Names: sugar pill
  Arms: Phase 1 -Placebo, Phase 2 -Placebo; Phase 1 -Placebo, Phase 2 -Ranolazine; Phase 1 -Ranolazine, Phase 2 -Placebo

SUMMARY:
The goal of this study is to evaluate whether supervised treadmill exercise combined with ranolazine 1000 mg twice daily provides an incremental benefit in absolute walking distance over supervised exercise alone in patients with stable claudication. Investigators also seek to determine if the administration of ranolazine provides a sustained benefit after the completion of a supervised exercise regimen. Lastly, investigators wish to determine whether both exercise and ranolazine improves peak oxygen consumption and anaerobic threshold in patients with stable claudication.

DETAILED DESCRIPTION:
The treatment groups are:

A. Group A will be randomized to a 12 week supervised exercise program and ranolazine, (Ranexa) 1000 mg orally, twice daily, by mouth.

B. Group B will be randomized to a 12 week supervised exercise program and placebo.

After the 12 week supervised exercise program, all participants will undergo a second randomization to ranolazine or placebo for an additional 12 weeks, during which independent walking will be encouraged.

Both groups will participate in a two week lead-in period after each randomization of the trial, allowing for the stabilization of their medications and dosing of ranolazine. Medications such as cilostazol, calcium channel blockers and nitrates will be discontinued during the lead-in period, unless their use is for management for high blood pressure. Anti-platelet (blood thinner) medications will be continued throughout the trial.

ELIGIBILITY:
Inclusion Criteria:

* Males or females greater than 40 years of age.
* Documented peripheral arterial disease
* Stable lower extremity intermittent claudication (Rutherford class 1-3) for 3 months.

Exclusion Criteria:

* Critical limb ischemia (Rutherford class 4-6).
* Percutaneous or surgical lower extremity revascularization within last 12 months.
* Myocardial infarction within the last 6 months.
* cardiac surgery within the last 6 months.
* Unstable angina
* Stable chronic angina
* New York Heart Association Class II-IV heart failure
* Left ventricular ejection fraction less than or equal to 35%
* Venous thromboembolism within the last 6 months.
* Uncontrolled high blood pressure, defined as systolic blood pressure greater than or equal to 180 mmHg or diastolic blood pressure greater than or equal to 110 mmHg.
* Allergy to ranolazine.
* corrected QT interval (QTc) greater than or equal to 440 ms in males or 460 ms in females.
* Pregnant or nursing females.
* Chronic dialysis therapy.
* Significant liver impairment (defined as transaminases greater than or equal to 3 times the upper limit of normal) within the last 6 months.
* Concomitant use of Cytochrome P450-3A (CYP3A) inhibitors
* Concomitant use of CYP3A inducers
* QTc prolonging agents
* Orthopedic or neurologic disorders that prevent treadmill walking.
* Current participation in a structured exercise program.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2009-05; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura Franny, M.D., Principal Investigator — Corewell Health East
Locations (1):
- William Beaumont Hospital, Royal Oak, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share individual participant data

RESULTS

PARTICIPANT FLOW:
Period: Phase 1
Arm/Group | Phase 1-Ranolazine, Phase 2-Ranolazine | Phase 1 -Ranolazine, Phase 2 -Placebo | Phase 1 -Placebo, Phase 2 -Ranolazine | Phase 1 -Placebo, Phase 2 -Placebo
Started | 7 | 6 | 8 | 8
Completed | 2 | 4 | 3 | 6
Not Completed | 5 | 2 | 5 | 2
Not completed — Physician Decision | 4 | 0 | 1 | 2
Not completed — Withdrawal by Subject | 0 | 2 | 4 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0
Period: Phase 2
Arm/Group | Phase 1-Ranolazine, Phase 2-Ranolazine | Phase 1 -Ranolazine, Phase 2 -Placebo | Phase 1 -Placebo, Phase 2 -Ranolazine | Phase 1 -Placebo, Phase 2 -Placebo
Started | 2 | 4 | 3 | 6
Completed | 1 | 4 | 2 | 6
Not Completed | 1 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Missing data for 4 participants in Ranolazine/Ranolazine group, and 2 participants in placebo/Ranolazine group.
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1-Ranolazine, Phase 2-Ranolazine | Phase 1 -Ranolazine, Phase 2 -Placebo | Phase 1 -Placebo, Phase 2 -Ranolazine | Phase 1 -Placebo, Phase 2 -Placebo | Total
Number analyzed (Participants) | 3 | 6 | 6 | 8 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 2 | 1 | 4 | 8
  >=65 years | 2 | 4 | 5 | 4 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.0 (3.6) | 69.7 (6.9) | 77.0 (10.5) | 65.8 (14.9) | 70.1 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 1 | 0 | 3
  Male | 3 | 4 | 5 | 8 | 20
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 6 | 6 | 8 | 23

OUTCOME MEASURES:

1. Primary Outcome: Percentage Increase in Absolute Walking Distance Following Phase 1
Description: Change in absolute walking distance in meters from baseline to 12 week follow-up treadmill test, as a percentage from baseline treadmill test
Time Frame: 12 weeks
Population: Missing data for 12 week test in 1 subject in Ranolazine/Ranolazine group, 1 subject in Ranolazine/placebo group, and 3 subjects in placebo/placebo group
Measure: Median (Inter-Quartile Range); unit: percentage of baseline
Arm/Group | Phase 1-Ranolazine, Phase 2-Ranolazine | Phase 1 -Ranolazine, Phase 2 -Placebo | Phase 1 -Placebo, Phase 2 -Ranolazine | Phase 1 -Placebo, Phase 2 -Placebo
Number analyzed (Participants) | 1 | 3 | 3 | 3
percentage of baseline | 112 [112 to 112] | 108 [105 to 121] | 145 [127 to 216] | 155 [142 to 166]

2. Secondary Outcome: Percentage Increase in Absolute Walking Distance Following Phase 2
Description: Change in absolute walking distance in meters from baseline to 24 week follow-up treadmill test, as a percentage from baseline treadmill test
Time Frame: 24 weeks
Population: Missing data from one subject 24 week treadmill test in placebo/placebo group
Measure: Median (Inter-Quartile Range); unit: percentage of baeline
Arm/Group | Phase 1-Ranolazine, Phase 2-Ranolazine | Phase 1 -Ranolazine, Phase 2 -Placebo | Phase 1 -Placebo, Phase 2 -Ranolazine | Phase 1 -Placebo, Phase 2 -Placebo
Number analyzed (Participants) | 1 | 4 | 2 | 5
percentage of baeline | 98 [98 to 98] | 120 [107 to 131] | 181 [163 to 200] | 145 [121 to 148]

ADVERSE EVENTS:
Time Frame: 28 weeks
Description: Only 8 adverse events were collected: death, unstable angina, ischemic ST depression > 2 mm during exercise training, myocardial infarction, cerebrovascular accident, ventricular arrhythmias (non-sustained ventricular tachycardia (VT), sustained VT, ventricular fibrillation), advanced heart block (Mobitz II or Type III heart block), and congestive heart failure (CHF) requiring hospitalization.
  Adverse events were collected for the 20 patients completing at least baseline testing in Phase 1.
Arm/Group | Phase 1-Ranolazine, Phase 2-Ranolazine | Phase 1 -Ranolazine, Phase 2 -Placebo | Phase 1 -Placebo, Phase 2 -Ranolazine | Phase 1 -Placebo, Phase 2 -Placebo
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/5 | 0/4 | 0/8
Serious Adverse Events (participants affected / at risk) | 1/3 | 0/5 | 0/4 | 0/8
Other Adverse Events (participants affected / at risk) | 0/3 | 0/5 | 0/4 | 0/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1-Ranolazine, Phase 2-Ranolazine (N=3) | Phase 1 -Ranolazine, Phase 2 -Placebo (N=5) | Phase 1 -Placebo, Phase 2 -Ranolazine (N=4) | Phase 1 -Placebo, Phase 2 -Placebo (N=8)
myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Early termination due to recruitment and retention difficulties, leading to small numbers of subjects. Missing data for several subjects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes